CLINICAL TRIAL: NCT02526641
Title: New AbbVie Direct Acting Antiviral (DAA) Treatment of Chronic Hepatitis C Infection - Effects on the Macrophage Activation Marker Soluble CD163, Portal Hypertension, and Metabolic Liver Function
Brief Title: Macrophages, Portal Hypertension, and Liver Function During AbbVie Treatment of Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: HCV sCD163 AbbVie
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis C
Keywords: Direct acting antiviral treatment; sCD163; Portal hypertension; Metabolic liver function; Cirrhosis
MeSH Terms: conditions — Hepatitis C; Hypertension, Portal; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AbbVie
  Interventions: Procedure: Functional Hepatic Nitrogen Clearance (FHNC); Procedure: Galactose Elimination Capacity (GEC); Procedure: Liver vein catheterization

INTERVENTIONS:
Procedure: Functional Hepatic Nitrogen Clearance (FHNC)
Procedure: Galactose Elimination Capacity (GEC)
Procedure: Liver vein catheterization

SUMMARY:
Investigation of the effects of the new Abbvie direct acting anti-viral (DAA) treatment of chronic viral hepatitis C infection on the macrophage specific activation marker soluble CD163, portal hypertension determined by the hepatic venous pressure gradient (HVPG), and metabolic liver function determined by the galactose elimination capacity (GEC) test and the functional hepatic nitrogen clearance (FHNC).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C genotype 1 or 4 patients initiating the new AbbVie treatment (paritaprevir, ritonavir, ombitasvir og dasabuvir sammen med ribavirin)
* Child-Pugh A liver cirrhosis

Exclusion Criteria:

* Severe liver dysfunction - Child-Pugh klasse B-C
* Life expectancy less than 6 months
* planned liver transplantation or TIPS procedure within 6 months
* non-compliance to treatment or study procedures
* allergy to the DAA drugs used (paritaprevir, ritonavir, ombitasvir, dasabuvir, and ribavirin)
* pregnancy or expected pregnancy during the study (anti-conception has to be used)
* breast feeding
* portal vein thrombosis
* liver cancer or other malignancies
* alcohol consumption

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C patients initiating direct-acting anti-viral therapy.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change in the hepatic venous pressure gradient determined by liver vein catheterization from baseline to 12 weeks | 12 weeks
Change in the hepatic venous pressure gradient determined by liver vein catheterization from baseline to 1 year | 1 year

SECONDARY OUTCOMES:
Changes in the levels of the macrophage specific activation marker sCD163 | Before, during and after treatment - 60 weeks
Changes in metabolic liver function determined by the galactose elimination capacity (GEC) test | After 12 weeks treatment
Changes in the functional hepatic nitrogen clearance (FHNC) | After 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Denmark